CLINICAL TRIAL: NCT04693559
Title: Assessment of Nanocrystalline Hydroxyapatite Versus Autogenous Bone Grafts : A Comparative Clinical Study in Alveolar Cleft Grafting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdullah Hashim Ahmed, MBBS, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AssiutU011270
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Alveolar Cleft
MeSH Terms: interventions — poly(2-hydroxyethyl methacrylate)-nanocrystalline hydroxyapatite

STUDY DESIGN:
Intervention Model Description: Patient will be randomized into to groups according to the surgical procedures performed as follow
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autogenous iliac bone graft (group A) (Other): autogenous iliac bone graft will be used to fill the alveolar defect
  Interventions: Procedure: secondary alveolar bone graft; Procedure: harvesting of the autogenous bone graft
- Nano crystalline Hydroxyapatite (group B) (Other): Nano crystalline Hydroxyapatite will be used to fill the alveolar defect
  Interventions: Procedure: secondary alveolar bone graft; Procedure: Nanocrystalline Hydroxyapatite

INTERVENTIONS:
Procedure: secondary alveolar bone graft — Under general anaesthesia, the soft tissue in the gingiva surrounding the alveolar cleft will injected with 0.5% lidocaine with 1:100,000 parts of epinephrine. At the alveolar cleft site, gingival sulcus incisions will made on both the sides of the cleft. The tissue will then elevated beneath the periosteum. The mucosa of the nasal floor and the oral mucosa will dissected. Next, the bone particles will implanted into the bone defect. The cleft site will closed without tension by advancement of the gingival flaps
Procedure: harvesting of the autogenous bone graft — osteotome and then cut into small bone granules. The bone granules will then carefully placed into a syringe and pressed to its densest state by pushing the plunger
  Arms: autogenous iliac bone graft (group A)
Procedure: Nanocrystalline Hydroxyapatite — Nanocrystalline Hydroxyapatite will be used to fill the alveolar defect
  Arms: Nano crystalline Hydroxyapatite (group B)

SUMMARY:
This work aims to evaluate Nanocrystalline Hydroxyapatite versus Autogenous bone grafts in alveolar cleft grafting

DETAILED DESCRIPTION:
Alveolar cleft is the most common congenital bone defect. Since its introduction in 1972, alveolar bone grafting (ABG) has been widely accepted to correct alveolar bone defect in most cleft centres.The purpose of ABG is to restore the dental arch continuity, stabilize the maxilla, close the oronasal fistulae, facilitate subsequent orthodontic treatment, enhance nasal symmetry, establish better oral hygiene, limit growth disturbances, etc . Autologous bone grafting is the gold standard for treating alveolar clefts, with the iliac crest , bone being the most widely accepted donor site(Tan, Brogan et al. 1996.New bone graft substitutes have been devised in recent decades, such as demineralized bone matrix (DBM), bone morphogenetic proteins (BMPs), calcium phosphate (CP), calcium sulfate (CS), hydroxyapatite (HA), highly purified bovine xenograft, and more, but clinical evidence of their efficacy varies among clinical and experimental studies [4] With the advent of new biomaterials, which may include or consist of allogenic bone source such as collagen membranes, hydroxyapatite crystals, tricalcium phosphate powder that has been increased consideration for their placement in the repair of alveolar clefts as well as other dental applications

ELIGIBILITY:
Inclusion Criteria:

* Age (7 - 12 years )
* Non-syndromic CLA or CLP
* More than 6 months of follow-up

Exclusion Criteria:

* History of previous alveolar surgery
* History of active infection or underlying disease such as hematologic disorders , neoplasm, and immune deficiency
* Patients who had received primary or tertiary ABG

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Measuring of bone volume 6 months post-operative | 6 months
  compare between outcome of nanocrystalline hydroxyapatite versus autogenous bone graft in alveolar bone grafting regarding the newly formed bone volume

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Boyne PJ, Sands NR. Secondary bone grafting of residual alveolar and palatal clefts. J Oral Surg. 1972 Feb;30(2):87-92. No abstract available. PMID 4550446
- [Background] Kyung H, Kang N. Management of Alveolar Cleft. Arch Craniofac Surg. 2015 Aug;16(2):49-52. doi: 10.7181/acfs.2015.16.2.49. Epub 2015 Aug 11. PMID 28913221
- [Background] Cypher TJ, Grossman JP. Biological principles of bone graft healing. J Foot Ankle Surg. 1996 Sep-Oct;35(5):413-7. doi: 10.1016/s1067-2516(96)80061-5. PMID 8915864
- [Background] Feinberg SE, Weisbrode SE, Heintschel G. Radiographic and histological analysis of tooth eruption through calcium phosphate ceramics in the cat. Arch Oral Biol. 1989;34(12):975-84. doi: 10.1016/0003-9969(89)90055-1. PMID 2558643
- [Background] Fernyhough JC, Schimandle JJ, Weigel MC, Edwards CC, Levine AM. Chronic donor site pain complicating bone graft harvesting from the posterior iliac crest for spinal fusion. Spine (Phila Pa 1976). 1992 Dec;17(12):1474-80. doi: 10.1097/00007632-199212000-00006. PMID 1471005
- [Background] Porter AE, Patel N, Skepper JN, Best SM, Bonfield W. Effect of sintered silicate-substituted hydroxyapatite on remodelling processes at the bone-implant interface. Biomaterials. 2004 Jul;25(16):3303-14. doi: 10.1016/j.biomaterials.2003.10.006. PMID 14980425
- [Background] Mankin HJ, Gebhardt MC, Jennings LC, Springfield DS, Tomford WW. Long-term results of allograft replacement in the management of bone tumors. Clin Orthop Relat Res. 1996 Mar;(324):86-97. doi: 10.1097/00003086-199603000-00011. PMID 8595781